CLINICAL TRIAL: NCT04773600
Title: A Phase 3, 4-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.15% Administered QD in Subjects With Atopic Dermatitis
Brief Title: Trial of PDE4 Inhibition With Roflumilast for the Management of Atopic Dermatitis (INTEGUMENT-II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-151-312
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Cream 0.15% (Experimental): Participants apply roflumilast cream 0.15% once daily (qd) for 4 weeks.
  Interventions: Drug: Roflumilast Cream
- Vehicle Cream (Placebo Comparator): Participants apply vehicle cream qd for 4 weeks.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Roflumilast Cream — Roflumilast cream 0.15% for topical application
  Other Names: ARQ-151
  Arms: Roflumilast Cream 0.15%
Drug: Vehicle cream — Vehicle cream for topical application
  Arms: Vehicle Cream

SUMMARY:
This study will assess the safety and efficacy of ARQ-151 cream vs vehicle applied once a day for 4 weeks by subjects with atopic dermatitis (eczema). This is a parallel group, double blind, vehicle-controlled study in which ARQ-151 0.15% cream or vehicle is applied once daily (qd) for 4 weeks by participants with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent and, if appropriate, assent as required by local laws.
2. Males and females, ages 6 years and older at time of signing Informed Consent (Screening). Only subjects 18 years and older will be enrolled at sites located in the province of Québec in Canada.
3. Diagnosed with atopic dermatitis 6 months duration (3 months for children), as determined by the Investigator. Stable disease for the past 4 weeks with no significant flares in atopic dermatitis before screening.
4. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline/Day 1. In addition, sexually active FOCBP must agree to use at least one form of a highly effective or barrier method of contraception throughout the trial.
5. In good health as judged by the Investigator.
6. Subjects considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

1. Subjects with any serious medical condition or clinically significant abnormality that would prevent study participation or place the subject at significant risk, as judged by the Investigator
2. Has unstable AD or any consistent requirement for high potency topical steroids.
3. Subjects who are unwilling to refrain from prolonged sun exposure and from using a tanning bed or other artificial light emitting devices (LEDs) for 4 weeks prior to Baseline/Day 1 and during the study.
4. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
5. Previous treatment with ARQ-151.
6. Subjects with a history of chronic alcohol or drug abuse within 6 months prior to Screening.
7. Parent(s)/legal guardian(s) who are unable to communicate, read, or understand the local language(s). Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
8. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects living in the same house.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (53):
- United States (44):
  - Arcutis Clinical Site 31, Birmingham, Alabama
  - Arcutis Clinical Site 51, Fort Smith, Arkansas
  - Arcutis Clinical Site 46, Inglewood, California
  - Arcutis Clinical Site 19, San Diego, California
  - Arcutis Clinical Site 36, San Diego, California
  - Arcutis Clinical Site 13, Santa Monica, California
  - Arcutis Clinical Site 54, Centennial, Colorado
  - Arcutis Clinical Site 55, Boca Raton, Florida
  - Arcutis Clinical Site 30, Coral Gables, Florida
  - Arcutis Clinical Site 37, Delray Beach, Florida
  - Arcutis Clinical Site 58, Miami, Florida
  - Arcutis Clinical Site 41, Miami, Florida
  - Arcutis Clinical Site 11, Sanford, Florida
  - Arcutis Clinical Site 57, West Palm Beach, Florida
  - Arcutis Clinical Site 62, Boise, Idaho
  - Clinical Site 04, Plainfield, Indiana
  - Arcutis Clinical Site 43, Louisville, Kentucky
  - Arcutis Clinical Site 63, Baton Rouge, Louisiana
  - Arcutis Clinical Site 42, Lake Charles, Louisiana
  - Arcutis Clinical Site 38, Mandeville, Louisiana
  - Arcutis Clinical Site 06, Metairie, Louisiana
  - Arcutis Clinical Site 34, Rockville, Maryland
  - Arcutis Clinical Site 29, Clinton Township, Michigan
  - Arcutis Clinical Site 21, Fort Gratiot, Michigan
  - Arcutis Clinical Site 61, Troy, Michigan
  - Arcutis Clinical Site 245, Saint Joseph, Missouri
  - Arcutis Clinical Site 53, New York, New York
  - Arcutis Clinical Site 39, Rochester, New York
  - Arcutis Clinical Site 33, Stony Brook, New York
  - Arcutis Clinical Site 01, High Point, North Carolina
  - Arcutis Clinical Site 24, Hershey, Pennsylvania
  - Arcutis Clinical Site 07, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 35, Charleston, South Carolina
  - Arcutis Clinical Site 18, Charleston, South Carolina
  - Arcutis Clinical Site 15, North Charleston, South Carolina
  - Clinical Site 05, Austin, Texas
  - Arcutis Clinical Site 03, College Station, Texas
  - Arcutis Clinical Site 59, Frisco, Texas
  - Arcutis Clinical Site 250, Grapevine, Texas
  - Arcutis Clinical Site 52, Pflugerville, Texas
  - Arcutis Clinical Site 02, San Antonio, Texas
  - Arcutis Clinical Site 32, Orem, Utah
  - Arcutis Clinical Site 22, Burke, Virginia
  - Arcutis Clinical Site 17, Norfolk, Virginia
- Canada (9):
  - Arcutis Clinical Site 12, Calgary, Alberta
  - Arcutis Clinical Site 09, Surrey, British Columbia
  - Arcutis Clinical Site 26, Winnipeg, Manitoba
  - Arcutis Clinical Site 20, Ajax, Ontario
  - Arcutis Clinical Site 23, London, Ontario
  - Arcutis Clinical Site 25, Toronto, Ontario
  - Arcutis Clinical Site 16, Waterloo, Ontario
  - Arcutis Clinical Site 08, Drummondville, Quebec
  - Arcutis Clinical Site 27, Québec, Quebec

REFERENCES:
- [Derived] Simpson EL, Eichenfield LF, Alonso-Llamazares J, Draelos ZD, Ferris LK, Forman SB, Gooderham M, Gonzalez ME, Hebert AA, Kircik LH, Lomaga M, Moore A, Papp KA, Prajapati VH, Hanna D, Snyder S, Krupa D, Burnett P, Almaraz E, Higham RC, Chu DH, Berk DR. Roflumilast Cream, 0.15%, for Atopic Dermatitis in Adults and Children: INTEGUMENT-1 and INTEGUMENT-2 Randomized Clinical Trials. JAMA Dermatol. 2024 Nov 1;160(11):1161-1170. doi: 10.1001/jamadermatol.2024.3121. PMID 39292443

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast Cream 0.15%: Participants applied roflumilast cream 0.15% qd for 4 weeks.
- Vehicle Cream: Participants applied vehicle cream qd for 4 weeks.
Period: Overall Study
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Started | 451 | 232
Completed | 410 | 211
Not Completed | 41 | 21
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Lost to Follow-up | 10 | 6
Not completed — Adverse Event | 8 | 2
Not completed — Lack of Efficacy | 2 | 3
Not completed — Noncompliance | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Caregiver Elected Other Therapy | 1 | 0
Not completed — Emergency Travel Out of Country | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream | Total
Number analyzed (Participants) | 451 | 232 | 683
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (19.60) | 26.2 (18.94) | 27.2 (19.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 143 | 395
  Male | 199 | 89 | 288
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 16 | 67
  Not Hispanic or Latino | 397 | 213 | 610
  Unknown or Not Reported | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 268 | 138 | 406
  Black or African-American | 96 | 50 | 146
  Asian | 51 | 30 | 81
  American-Indian or Alaska Native | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Multiple | 12 | 8 | 20
  Other | 19 | 5 | 24
Randomization validated Investigator Global Assessment for Atopic Dermatitis (vIGA) Baseline Score [Count of Participants; unit: Participants] — vIGA-AD is a 5-point scale assessing the severity of AD, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity. This is the baseline vIGA entered into the IWRS used for randomization.
  Participants
    Mild | 109 | 53 | 162
    Moderate | 342 | 179 | 521
Investigator-Verified vIGA Baseline Score [Count of Participants; unit: Participants] — vIGA-AD is a 5-point scale assessing the severity of AD, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity. This is the baseline vIGA data that have undergone data verification by the investigator.
  Participants
    Mild | 108 | 53 | 161
    Moderate | 343 | 179 | 522
WI-NRS Baseline Score ≥4 [Count of Participants; unit: Participants] — The number of participants with average, weekly baseline WI-NRS score ≥4 is presented. WI-NRS is a subject-reported severity of itch at its highest intensity during the previous 24-hour period. The scale is from '0 to 10' ("no itch" to "worst imaginable itch"), with higher scores indicating greater symptom severity.
  Participants
    ≥4 | 359 | 181 | 540
    ≤3 | 92 | 51 | 143
Baseline Eczema Area and Severity Index (EASI) Score [Median (Inter-Quartile Range); unit: units on a scale] — EASI is an instrument to measure the severity and extent of AD. The body is first divided into 4 areas: head (10% of skin), arms (20%), trunk (30%), and legs (40%). Then, the area affected is scored from 0 (0% involvement) to 6 (90-100% involvement), and severity is scored from 0 ('none') to 3 ('severe'). EASI combines the area affected and severity ratings to get a final composite score ranging from 0 (no disease) to 72 (maximal disease). Note that palms and soles were treated as appropriate but were not counted towards any measurements of EASI.
  units on a scale | 8.50 [6.2 to 12.3] | 8.4 [6.45 to 12.00] | 8.50 [6.40 to 12.20]

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Success at Week 4
Description: The percentage of participants achieving viGA-AD "success" is presented with multiple imputation of missing observations. viGA-AD "success" is defined as a viGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from Baseline. The viGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4 where 0 is clear), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 28.9 | 12.0
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA Success at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.962 to 5.183] — Stratified by pooled study site and vIGA-AD randomization strata

2. Secondary Outcome: Achievement of vIGA-AD Success at Week 4 in Participants With "Moderate" Baseline Scores
Description: The percentage of participants with moderate baseline scores achieving viGA-AD "success" is presented with multiple imputation of missing observations. viGA-AD "success" is defined as a viGA-AD score of 'clear' or 'almost clear' PLUS a 2-grade improvement from baseline in participants with a 'moderate' baseline viGA-AD score. The viGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants who were included in the "moderate" baseline vIGA-AD group during randomization are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 342 | 179
percentage of participants | 32.9 | 13.1
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA Success at Week 4 in Participants with Baseline vIGA = 'Moderate'; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site; Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.996 to 5.687] — Stratified by pooled study site

3. Secondary Outcome: vIGA-AD Success at Week 2
Description: as for outcome 1
Time Frame: Week 2
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 17.7 | 5.3
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Success at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 4.42, 95% CI 2-sided [2.281 to 8.658] — Stratified by pooled study site and vIGA-AD randomization strata

4. Secondary Outcome: vIGA-AD Success at Week 1
Description: as for outcome 1
Time Frame: Week 1
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 5.9 | 3.1
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Success at Week 1; Test type: Superiority; p = 0.1156, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.832 to 4.782] — Stratified by pooled study site and vIGA-AD randomization strata

5. Secondary Outcome: Achievement of a 4-point Reduction at Week 4 in the Average, Weekly Worst Itch Numeric Rating Scale (WI-NRS) in Participants With Baseline WI-NRS Score ≥4
Description: The percentage of participants with a baseline WI-NRS ≥ 4 achieving WI-NRS success is presented with multiple imputation of missing observations. The WI-NRS is a simple, single item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the previous 24 hours (higher scores indicate higher itch severity).
Time Frame: Week 4
Population: All randomized participants who were ≥12 years of age, had an average weekly WI-NRS pruritus score ≥4 at baseline, and completed at least 4 of 7 evaluable daily WI-NRS questionnaires during the last 7 days of the Screening period are included. Multiple imputation was used to handle missing cases.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 264 | 136
percentage of participants | 30.2 [24.77 to 36.31] | 12.4 [7.77 to 19.26]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; ≥4-Point Reduction in WI-NRS at Week 4; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.448 to 5.066] — Stratified by pooled study site and vIGA-AD randomization strata

6. Secondary Outcome: Achievement of a 4-point Reduction at Week 2 in the WI-NRS in Participants With Baseline WI-NRS Score ≥4
Description: as for outcome 5
Time Frame: Week 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 264 | 136
percentage of participants | 22.3 [17.66 to 27.82] | 6.9 [3.66 to 12.56]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; ≥4-Point Reduction in WI-NRS at Week 2; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 3.55, 95% CI 2-sided [1.591 to 7.927] — Stratified by pooled study site and vIGA-AD randomization strata

7. Secondary Outcome: Achievement of a 4-point Reduction at Week 1 in the WI-NRS in Participants With Baseline WI-NRS Score ≥4
Description: as for outcome 5
Time Frame: Week 1
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 264 | 136
percentage of participants | 11.2 [7.89 to 15.57] | 1.6 [0.44 to 5.58]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; ≥4-Point Reduction in WI-NRS at Week 1; Test type: Superiority; p = 0.0020, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 7.84, 95% CI 2-sided [1.717 to 35.764] — Stratified by pooled study site and vIGA-AD randomization strata

8. Secondary Outcome: Achievement of ≥75% Decrease From Baseline at Week 4 in the Eczema Area and Severity Index (EASI-75)
Description: The percentage of participants achieving EASI-75 is presented with multiple imputation of missing observations. EASI-75 is a ~75% reduction from the baseline EASI score. EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum = of the severity rating (0 to 3 with 3 being the most severe) for four clinical signs are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 42.0 [37.45 to 46.72] | 19.7 [15.04 to 25.44]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; EASI-75 at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 3.23, 95% CI 2-sided [2.108 to 4.964] — Stratified by pooled study site and vIGA-AD randomization strata

9. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 4
Description: The percentage of participants scoring 'clear' or 'almost clear' on viGA-AD is presented with multiple imputation of missing observations. The viGA-AD is a static evaluation of qualitative overall AD severity. This global assessment scale is an ordinal scale with five severity grades (0 'clear' to 4 'severe'), with higher scores indicative of greater symptom severity.
Time Frame: Week 4
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 39.0 | 16.9
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 4; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 3.39, 95% CI 2-sided [2.191 to 5.240] — Stratified by pooled study site and vIGA-AD randomization strata

10. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 2
Description: as for outcome 9
Time Frame: Week 2
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 27.6 | 10.7
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 2; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 3.50, 95% CI 2-sided [2.097 to 5.854] — Stratified by pooled study site and vIGA-AD randomization strata

11. Secondary Outcome: Achievement of vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 1
Description: as for outcome 9
Time Frame: Week 1
Population: All randomized participants are included.
Measure: Number; unit: percentage of participants
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
Number analyzed (Participants) | 451 | 232
percentage of participants | 14.2 | 6.2
Statistical Analysis 1: Comparison: Roflumilast Cream 0.15% vs Vehicle Cream; vIGA-AD Score of 'Clear' or 'Almost Clear' at Week 1; Test type: Superiority; p = 0.0050, Cochran-Mantel-Haenszel; Stratified by pooled study site and vIGA-AD randomization strata; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.312 to 4.993] — Stratified by pooled study site and vIGA-AD randomization strata

ADVERSE EVENTS:
Time Frame: Up to ~29 days
Description: All randomized participants who received ≥1 dose of study intervention are included, according to actual treatment received. Note that 1 participant was randomized to vehicle but did not receive ≥1 dose of study treatment; one additional participant was randomized to vehicle but instead received active roflumilast.
Arm/Group | Roflumilast Cream 0.15% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/452 | 0/232
Serious Adverse Events (participants affected / at risk) | 4/452 | 0/232
Other Adverse Events (participants affected / at risk) | 0/452 | 0/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.15% (N=452) | Vehicle Cream (N=232)
Nerve compression (Injury, poisoning and procedural complications) | 1 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT04773600/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04773600/SAP_001.pdf